CLINICAL TRIAL: NCT07384416
Title: QL1706 Combined With Lenvatinib and Nab-Paclitaxel in the Treatment of Recurrent or Refractory Advanced Penile Cancer: a Single Arm, Phase II Study
Brief Title: Single-Arm Trial of QL1706, Lenvatinib, and Nab-Paclitaxel for Advanced Refractory Penile Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-740-01
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Penile Cancer
MeSH Terms: conditions — Penile Neoplasms | interventions — lenvatinib; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: QL1706 + Lenvatinib + Nab-Paclitaxel

INTERVENTIONS:
Drug: QL1706 + Lenvatinib + Nab-Paclitaxel — Lenvatinib: 8 mg once daily (for body weight <60 kg) or 12 mg once daily (for body weight ≥60 kg).
  QL1706: 5 mg/kg, administered by intravenous infusion (iv) on Day 1 of each cycle.
  Nab-Paclitaxel: 260 mg/m², administered by intravenous infusion (iv) on Day 1 of each cycle.
  Treatment Cycle: Each cycle is 21 days. The combination therapy will be administered for 4 cycles.
  Maintenance Therapy:
  QL1706 treatment will continue for up to 1 year. Lenvatinib will be taken orally until disease progression.

SUMMARY:
The aim of this clinical trial is to evaluate the combination of QL1706, Lenvatinib, and Nab-Paclitaxel for the treatment of recurrent or refractory advanced penile cancer and to assess the safety of this regimen. The main questions it aims to answer are:

* Can the combination of QL1706, Lenvatinib, and Nab-Paclitaxel shrink tumors or prolong the time to disease progression in participants with advanced penile cancer?
* What side effects do participants experience while taking this three-drug combination?

Researchers will compare the tumor response in participants receiving this treatment with historical data from standard therapies to determine whether the new combination is more effective for this type of cancer. This is a single-arm study, meaning all participants will receive the same investigational combination.

Participants will:

* Receive intravenous infusions of QL1706 and Nab-Paclitaxel every 21 days, along with daily oral Lenvatinib capsules.
* Continue treatment cycles until disease progression, unacceptable side effects occur, or they choose to withdraw from the study.
* Attend regular clinic visits for imaging scans (such as CT scans), physical examinations, and blood tests to monitor treatment response and safety.
* Have their tumors measured by scans at scheduled intervals to evaluate treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Histologically or cytologically confirmed penile squamous cell carcinoma.
3. Previous treatment with chemotherapy, immunotherapy, and/or targeted therapy.
4. At least one measurable target lesion according to RECIST 1.1 criteria.
5. ECOG performance status score of ≤ 2.
6. Adequate bone marrow function: Hemoglobin (Hb) ≥ 75 g/L, White Blood Cell count (WBC) ≥ 3.0×10⁹/L, Absolute Neutrophil Count (ANC) ≥ 1.5×10⁹/L, Platelet count (PLT) ≥ 100×10⁹/L.
7. Adequate organ function:

   Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), and Alkaline Phosphatase (ALP) ≤ 2.5 times the upper limit of normal (ULN); Total bilirubin ≤ 1.5 × ULN.

   Serum creatinine ≤ 1.5 × ULN.
8. Life expectancy of ≥ 12 months.
9. No significant history of severe cardiac, pulmonary, hepatic, or other major organ diseases.
10. The patient understands the study procedures and provides written informed consent to participate in the study.

Exclusion Criteria:

1. Participation in any investigational drug study within 4 weeks prior to the start of treatment.
2. Concurrent active cancer other than penile squamous cell carcinoma, or a history of other malignancies within the past 5 years, except for the following:

   * (1) Cured non-melanoma skin cancer;
   * (2) Incidentally discovered, low-risk, and curative tumors, including but not limited to low-risk prostate cancer (T1a, Gleason score <6, PSA <0.5 ng/ml) and superficial bladder cancer;
   * (3) Other solid tumors that have undergone curative treatment with no evidence of recurrence or metastasis for 5 years or more.
3. Other serious, poorly controlled concurrent illnesses that may be aggravated by the combination therapy, including but not limited to:

   * (1) History of severe or acute exacerbation within the past 6 months involving the cardiovascular, hepatic, respiratory, renal, hematological, endocrine, or neuropsychiatric systems;
   * (2) Active infection requiring antibiotic treatment within 2 weeks prior to enrollment;
   * (3) Congestive heart failure (Class III-IV);
   * (4) Unstable angina or myocardial infarction within the past 6 months;
   * (5) Untreated active Hepatitis B virus (HBV) infection. *Note: Subjects with HBV meeting the following criteria are eligible: HBV viral load must be <1000 copies/ml (200 IU/ml) before the first dose, and the subject must receive anti-HBV therapy throughout the study treatment period to prevent reactivation. Subjects who are anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-) do not require prophylactic anti-HBV therapy but require close monitoring for reactivation.*
   * (6) Active Hepatitis C virus (HCV) infection (HCV antibody positive and HCV-RNA level above the limit of detection).
4. Administration of a live vaccine within 30 days prior to the first dose (Cycle 1, Day 1). *Inactivated seasonal influenza vaccines administered by injection are permitted within 30 days prior to the first dose; however, live attenuated influenza vaccines administered intranasally are not permitted.*
5. Diagnosis of immunodeficiency or receipt of systemic corticosteroid therapy (>10 mg/day prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first study dose. *Physiologic doses of corticosteroids (≤10 mg/day prednisone or equivalent) are permitted.*
6. History of Human Immunodeficiency Virus (HIV) infection (i.e., positive HIV1/2 antibody test).
7. Systemic treatment with Chinese herbal medicines with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use to control pleural effusion) within 2 weeks prior to enrollment.
8. Active autoimmune disease that has required systemic treatment (e.g., with disease-modifying agents, corticosteroids, or immunosuppressants) within the past 2 years.
9. Any other history, disease, concurrent condition, therapy, or laboratory abnormality that, in the investigator's judgment, might compromise the results, interfere with the subject's full participation throughout the study, or make the subject unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free Survival） | 2 year

SECONDARY OUTCOMES:
ORR (Objective Response Rate） | week 12